CLINICAL TRIAL: NCT06695429
Title: Suplementación Con Zumo de REmolacha Para Prevenir la Nefropatía Asociada a Contraste Durante la hospitalización Por Síndrome Coronario Agudo Sin elevación Del ST
Brief Title: Supplementation With Beetroot Juice to Prevent Contrast Associated Nephropathy During Hospitalization for Acute Coronary Syndrome Without ST Elevation
Acronym: RENACS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario Santa Lucia (Other)
Responsible Party: Principal Investigator, Jose Manuel Andreu Cayuelas, Principal Investigator, Hospital General Universitario Santa Lucia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RENACS
Record Dates: First submitted 2024-10-14; First posted 2024-11-19 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Non ST Segment Elevation Acute Coronary Syndrome; Contrast Induced Nephropathy
Keywords: Beetroot juice; Inorganic nitrates; Contrast induced nephropathy; Non ST elevation acute coronary syndrome; Percutaneous coronary intervention; Contrast

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Beetroot juice supplementation (Experimental): Supplementation with 500 mL of beetroot juice daily in 2 doses of 250 mL, for 7 days, or until hospital discharge, and a recommendation to maintain a diet rich in vegetables with high nitrate content after discharge.
  (In addition to usual treatment with hydration and statins to prevent contrast induced nephropathy)
  Interventions: Dietary Supplement: Beetroot juice
- Usual care (No Intervention): Usual treatment with hydration and statins to prevent contrast induced nephropathy

INTERVENTIONS:
Dietary Supplement: Beetroot juice — Supplementation with 500 mL of beetroot juice daily in 2 doses of 250 mL, for 7 days, or until hospital discharge, and a recommendation to maintain a diet rich in vegetables with high nitrate content after discharge.
  Arms: Beetroot juice supplementation

SUMMARY:
The goal of this study is to compare the possible beneficial effect of beetroot juice supplementation versus the usual management during hospitalization to prevent contrast-induced nephropathy after cardiac catheterizations.

The study includes patients diagnosed with non-ST elevation acute coronary syndrome with a possible indication for catheterism and high risk of kidney injury related to iodinated contrast.

The intervention group will drink 500 mL (2 glasses daily, at breakfast and dinner) of beetroot juice added to the usual diet for 7 days or until hospital discharge and will receive the recommendation to maintain a diet rich in inorganic nitrates. The control group will receive the usual diet and recommendations. In both cases, other therapies will be prescribed to prevent contrast-induced nephropathy (hydration and statins) if there is no contraindication.

Our hypothesis is that a compound present in beetroot juice, inorganic nitrates, can prevent the deterioration of kidney function related to contrast due to its vasodilatory effect, in addition to improving the subsequent prognosis of coronary heart disease due to its anti-inflammatory and antiproliferative effects, protector of the endothelium and inhibitor of platelet aggregation. Beetroot juice could also be beneficial in this context due to the antioxidant effect of the betalains it contains.

DETAILED DESCRIPTION:
Contrast-induced nephropathy (CIN) is a common complication in patients admitted for acute coronary syndrome (ACS) who undergo percutaneous coronary intervention (PCI).

Although the deterioration of renal function is generally reversible, avoiding CIN is of great importance as it is associated with worse prognosis, including greater need for renal replacement therapies and greater mortality.

Inorganic nitrates (NO3-) are the most promising therapy to prevent CIN, due to their ability to be metabolized to nitric oxide (NO), whose vasodilator effect protects renal perfusion. In addition, NO has other potential benefits in ACS due to its anti-inflammatory, antiproliferative, endothelium protective, and platelet aggregation inhibitor effects.

The recent NITRATE-CIN study has shown that the administration of 12 mmol/24 h of KNO3 for 5 days to patients admitted for non-ST elevation (NSTE) ACS undergoing PCI not only significantly reduced the risk of CIN, but also prevented the deterioration of kidney function and significantly reduced major cardiovascular complications (MACE) during follow-up.

However, there is currently no comercially available presentation for KNO3 and its administration could be associated with hyperkalemia.

Furthermore, evidence of its use during admission for NSTE ACS comes from a single-center study with a small representation of Mediterranean population, which raises doubts about the validity of these results in our patients.

Drinking beetroot juice is a very promising alternative to administer NO3- during admission for NSTE ACS, due to its greater availability, simplicity of administration and minor risk of adverse effects such as hyperkalemia.

500 mL of beetroot juice daily contain approximately 11 mmol of NO3-, their consumption increases plasma NO similar to KNO3 and, in patients with chronic coronary syndrome, has been shown to reduce the risk of stent restenosis and MACE during follow-up, without significant adverse effects.

Objetives:

* Describe the effect of dietary supplementation with beetroot juice during hospital admission for NSTE ACS in the prevention of CIN after PCI.
* Assess the tolerance of beetroot juice supplementation during admission by NSTE ACS and its possible relationship with adverse effects such as hyperkalemia.
* Analyze the effect of the administration of beetroot juice during admission and recommendation upon discharge to maintain a diet rich in vegetables with a high content of nitrates on renal function during follow-up, including the need for initiation of renal replacement therapies.
* Evaluate the relationship between the effect of the administration of beetroot juice during hospitalization and the recommendation upon discharge to maintain a diet rich in vegetables with high nitrate content with MACE during the first year of follow-up after NSTE ACS.

Study design:

PROBE study (Prospective Randomized Open, Blinded End-point) Nutritional intervention study. Unicentric. Study population: Patients >18 years old who enter our center with a diagnosis ofNSTE-ACS with indication for PCI and moderate or high risk of CIN (Mehran scale score not including contrast ≥ 6).

Intervention: Supplementation with 500 mL of beetroot juice daily in 2 doses of 250 mL, for 7 days or until discharge from admission for NSTE-ACS. Recommendation to maintain a diet rich in vegetables with high nitrate content after discharge.

The control group will follow the usual management and diet. In both groups, it will be administered treatment with hydration and statins to prevent CIN.

Analyzed Variables:

Relationship between supplementation with 500 mL of beetroot juice daily during admission for NSTE-ACS with:

* Incidence of CIN during admission according to KDIGO creatinine criteria (increased Serum creatinine ≥0.3 mg/dL in the first 48 hours or ≥1.5 times the baseline value during the week after PCI)
* Incidence of dropout due to juice intolerance in the intervention group, hyperkalemia (defined as K>5.5 mEq/L with previous normal values) or others adverse events during admission.
* Evolution of glomerular filtration rate and need for renal replacement therapy during the first year after PCI.
* Incidence of MACE and total mortality during the first year after PCI. Personal history, characteristics of NSTEA CS and PCI and creatinine values at admission, after PCI, during follow-up and treatments administered values will also be registered.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Acute Coronary Syndrome without persistent ST segment elevation, with recommendation for invasive management according to the actual Clinical practice guidelines
* At least moderate or high risk of nephropathy associated with iodinated contrast (Mehran score (without including contrast volume) ≥ 6).

Exclusion Criteria:

* <18 years old or without capacity to give consent.
* Refusal to participate in the study.
* Known hypersensitivity to beetroot or any of its allergens.
* Pregnant.
* Inability to take food orally
* Serious illnesses (not related to ACS or kidney failure), which limits their life expectancy to a period predictably less than 1 year.
* On dialysis or predialysis at the time of inclusion.
* ACS with persistent ST segment elevation before inclusion.
* Shock or inotrope dependence at the time of inclusion
* PCI already performed before inclusion.
* Patients receiving intravenous nitroglycerin for > 1 hour before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Contrast-induced nephropathy | 7 days
  Defined as an increase in serum creatinine ≥0.3 mg/dL in the first 48 hours or ≥1.5 times the baseline value during the week after the first PCI performed on admission

SECONDARY OUTCOMES:
Number of Participants with In-hospital MACE (Major adverse cardiovascular events) | Up to 30 days
  Mortality from any cause, Myocardial infarction, PCI with unscheduled revascularization
Number of Participants with In-hospital hyperkalemia | Up to 30 days
  K >5.5 mEq/L (with previously normal values at admission)
Rate of Drop-out from beetroot juice during hospitalization | 7 days
  Abandonment of beetroot juice supplementation upon patient's request after having started it
Relative and absolute changes from baseline of serum creatinine and estimated glomerular filtration rate during follow-up | 1 year
  Change (Absolute and in porcentage from baseline) in serum creatinine (mg/mL) and glomerular filtration rate (estimated by CKD-EPI formula, in mL/min/1.73 m2) at 3-6 months and 9-12 months after PCI.
Number of Participants with Need for renal replacement therapy | 1 year
  Initiation of renal replacement therapy (Dialysis or Kidney transplant) during the follow-up.
Number of Participants with MACE during follow-up | 1 year
  Mortality from any cause, Myocardial infarction, PCI with unscheduled revascularization) during the first year after PCI

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Santa Lucía, Cartagena, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: ICF
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: At request from other investigators, contacting with the contact-author. To perform meta-analyses or future studies about this matter.